CLINICAL TRIAL: NCT05107687
Title: The Effectiveness of a Structured Smoking Cessation Program Versus Unassisted Smoking Cessation Methods in Cancer Patients Managed in a Community Health System
Brief Title: Effectiveness of Smoking Cessation Program in a Community Health System
Status: Enrolling by invitation | Type: Observational
Sponsor: Virtua Health, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-2021-02
Record Dates: First submitted 2021-10-05; First posted 2021-11-04 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assisted Smoking Cessation: Subject participates in a structured smoking cessation program hosted at Virtua Health which may be either smoking cessation group sessions or individual sessions and/or both. All participants will be provided with a list of smoking cessation resources.
  Description of Group Smoking Education and Support: These sessions are led by a Tobacco Treatment Specialist and include 2-3 sessions in-person or virtually and cover the following topics: Biological changes caused by nicotine, addiction, tips to quit smoking, health benefits to quitting smoking, types of nicotine replacement therapy, e-cigarettes and devices, aromatherapy, meditation and various resources. In addition, access to nicotine replacement therapies is optional.
  Interventions: Behavioral: Smoking cessation
- Unassisted Smoking Cessation: The subject receives no professional support but is provided with a list of smoking cessation resources, in this cohort the subject engages in smoking cessation with no assistance from a provider.
  Interventions: Behavioral: Smoking cessation

INTERVENTIONS:
Behavioral: Smoking cessation — Assisted Smoking Cessation- Subject is provided professional support provided by tobacco cessation specialist.
  Unassisted Smoking Cessation- Subject provided resources and attempts to quit smoking without professional support.
  The subject selects their preferred intervention.

SUMMARY:
Research efforts are needed to increase tobacco cessation support and to improve tobacco cessation efficacy. In addition, strategies must be identified to increase access to smoking cessation support and to develop processes to integrate smoking cessation into treatment plans for cancer patients.

DETAILED DESCRIPTION:
The Cancer Patient Tobacco Questionnaire (C-TUQ) survey tool will be used to address the primary and secondary outcome measures. This tool is publicly available on the National Cancer Institutes Grid-Enabled Measures website and was developed by NCI and the American Association for Cancer Research. This tool is a 22-item self-report survey designed to capture information about tobacco use by cancer patients and cancer survivors. Comparisons will be made for those patients that enroll in the structured smoking cessation program versus those patients that have opted to quit on their own.

Primary:

To determine the effectiveness of an intensive structured smoking cessation program (education and support) provided by a tobacco cessation trained specialist versus unassisted smoking cessation quitting methods (no support, patients have opted to stop on their own) in cancer patients seen in a community health care system

Secondary:

* Self-reported 7-day point-prevalence smoking abstinence at 6-month follow-up in patients participating in a structured smoking cessation program versus those patients that have quit smoking with professional support
* Self-reported 7-day point-prevalence smoking abstinence at 12-month follow-up in patients participating in a structured smoking cessation program versus those patients that have quit smoking without professional support, participants choosing to stop smoking on their own.
* Examine the impact of implementing a system level smoking cessation program into the ongoing management of our cancer patients who smoke.

ELIGIBILITY:
Inclusion Criteria:

Any Gender

* Over 18 years of age
* Able to read and understand English
* Able to sign the informed consent form
* A current cigarette smoker defined as smoking within 30 days
* Diagnosed with cancer and wants to quit smoking

Exclusion Criteria:

* • Individuals with Dementia

  * ECOG Performance Status 3-4
  * Survival prognosis less than 12 months
  * Currently participating in a smoking cessation program that is not provided by Virtua
  * Individuals who do not want to quit smoking
  * Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cancer patients who are actively smoking receiving treatment for any type of cancer, for patients who have completed treatment and cancer survivors.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Effectiveness of a Structured Smoking Cessation Program versus Unassisted Smoking Cessation Methods in Cancer Patients Managed in a Community Health System | 6 and 12 month intervals
  To determine the effectiveness of an intensive structured smoking cessation program versus unassisted smoking cessation quitting methods in cancer patients seen in a community health care system

SECONDARY OUTCOMES:
The Effectiveness of a Structured Smoking Cessation Program in Cancer Patients in a Community Health System The Effectiveness of a Structured Smoking Cessation Program versus Unassisted Smoking Cessatio | 6 and 12 month intervals
  * Self-reported 7-day point-prevalence smoking abstinence at 6-month follow-up in patients participating in a structured smoking cessation program versus those patients that have quit smoking without professional support.
  * Self-reported 7-day point-prevalence smoking abstinence at 12-month follow-up in patients participating in a structured smoking cessation program versus those patients that have quit smoking without professional support.
  * Examine the impact of implementing a system level smoking cessation program into the ongoing management of our cancer patients who smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Carducci, MSN, RN, CCRP, Principal Investigator — Virtua Health
Locations (1):
- Virtua Health, Voorhees Township, New Jersey, United States